CLINICAL TRIAL: NCT02499757
Title: Does Sweet Taste Potentiate Nicotine Cue Reactivity?
Acronym: FNC-nicotine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 1408014434; P50DA036151 (NIH)
Record Dates: First submitted 2014-10-24; First posted 2015-07-16 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Healthy
Keywords: Perception; brain response; nicotine; taste
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- flavor and sweetener (Experimental): E-cigarette with a novel flavor and sweetener added
  Interventions: Device: flavor and sweetener
- flavor and nicotine (Experimental): E-cigarette with a novel flavor and 12 mg nicotine added
  Interventions: Device: flavor and nicotine
- flavor, nicotine and sweetener (Experimental): E-cigarette with a novel flavor, sweetener, and 12 mg nicotine added
  Interventions: Device: flavor, nicotine and sweetener
- flavor (Experimental): E-cigarette with a novel flavor: without a sweetener and 12 mg nicotine added
  Interventions: Device: flavor

INTERVENTIONS:
Device: flavor and sweetener — maltol added as sweetener to e-cigarette with flavor
  Arms: flavor and sweetener
Device: flavor and nicotine — 12 mg of nicotine added to e-cigarette with flavor
  Arms: flavor and nicotine
Device: flavor, nicotine and sweetener — 12 mg nicotine and maltol (sweetener) added to e-cigarette with flavor
  Arms: flavor, nicotine and sweetener
Device: flavor — flavored e-cigarette stand alone without added nicotine and maltol (sweetener)
  Arms: flavor

SUMMARY:
The investigators' aim is to test the prediction that sweet taste perception enhances the ability of nicotine to induce neural plastic changes in brain reward circuits to increase the saliency, liking and brain reactivity to the sight and vaporized flavor of electronic cigarettes (e-cigarettes).

DETAILED DESCRIPTION:
Alternative tobacco products are becoming increasingly available in the US market and are promoted as potentially less deleterious compared to cigarettes. These products are increasing in usage as either a substitution for cigarette smoking or in addition to smoking. One particular appeal is that they often combine nicotine with sweet taste and flavors, which are themselves reinforcing. The primary goal of this project is to determine if sweet taste can potentiate the reinforcing properties of nicotine. Similar to nicotine, cues predicting the availability of carbohydrates can stimulate intake, even in the absence of hunger. The investigators have developed a novel flavor-nutrient conditioning paradigm to study the reinforcing properties of carbohydrates. Novel flavors are paired with 0 or 113 kcal carbohydrate and increases in flavor-cue reactivity (change in liking and brain response) when later sampled in the absence of the carbohydrate provide a measure of the reinforcing potency. For smokers, the aroma of tobacco is a potent cue that can promote smoking behavior. Using a modified version of our conditioning paradigm, our specific aim is to test the prediction that sweet taste perception enhances the ability of nicotine to induce neural plastic changes in brain reward circuits to increase the saliency, liking and brain reactivity to the sight and vaporized flavor of electronic cigarettes (e-cigarettes). Participants will smoke e-cigarettes that contain nicotine and an unsweetened vaporized flavor, nicotine and a sweet vaporized flavor or only a sweet vaporized flavor (no nicotine). The investigators predict that response in the nucleus accumbens and hypothalamus to the sight and vaporized flavor of the e-cigarette that was paired with nicotine and sweet taste will be greater than the responses to the sight and vaporized flavors associated with the other e-cigarettes. The investigators further predict that liking and wanting will increase more for the sight and vaporized flavor associated with both nicotine and sweet taste. This finding would provide strong evidence that sweet taste potentiates the reinforcement potency of nicotine and could therefore promote use.

ELIGIBILITY:
Inclusion Criteria:

* right handed
* non-daily smoker
* english speaking

Exclusion Criteria:

* serious or unstable medical illness (e.g., cancer);
* past or current history of alcoholism or consistent drug use;
* current and history of major psychiatric illness as defined by the DSM-IV criteria including eating disorders,
* medications that affect alertness (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, etc.) and any psychoactive drugs or anti-obesity agents;
* history of major head trauma with loss of consciousness;
* ongoing pregnancy;
* known taste or smell dysfunction;
* a diagnosis of diabetes;
* any known allergies or sensitivity, including to food, vapors or odors;
* pregnant or nursing women,
* history of metalworking, injury with shrapnel or metal slivers, and major surgery;
* history of pacemaker or neurostimulator implantation m) asthma, chronic obstructive pulmonary disease, bronchitis or any other lung disease.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on Rating: Liking | 2 days
  At baseline and 2 days post exposure, subjects will rate 'liking' using the general Labeled Hedonic Scale (LHS). The LHS is a vertical line scale with quasi-logarithmic spaced, with the label 'most imaginable dislike' in the bottom to 'most imaginable like' in the top, with the label 'neutral' in the middle (recoded to range of -100 to +100).

SECONDARY OUTCOMES:
percent signal change of nucleus accumbens from fMRI | on average 2 weeks
  brain response in nucleus accumbens and hypothalamus (in percent signal

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Small, Principal Investigator — The John B. Pierce Laboratory
Locations (1):
- The John B Pierce Laboratory, New Haven, Connecticut, United States

REFERENCES:
- [Background] Backinger CL, Fagan P, O'Connell ME, Grana R, Lawrence D, Bishop JA, Gibson JT. Use of other tobacco products among U.S. adult cigarette smokers: prevalence, trends and correlates. Addict Behav. 2008 Mar;33(3):472-89. doi: 10.1016/j.addbeh.2007.10.009. Epub 2007 Nov 4. PMID 18053653
- [Background] Drummond MB, Upson D. Electronic cigarettes. Potential harms and benefits. Ann Am Thorac Soc. 2014 Feb;11(2):236-42. doi: 10.1513/AnnalsATS.201311-391FR. PMID 24575993
- [Background] Fedoroff IC, Polivy J, Herman CP. The effect of pre-exposure to food cues on the eating behavior of restrained and unrestrained eaters. Appetite. 1997 Feb;28(1):33-47. doi: 10.1006/appe.1996.0057. PMID 9134093
- [Background] de Araujo IE, Lin T, Veldhuizen MG, Small DM. Metabolic regulation of brain response to food cues. Curr Biol. 2013 May 20;23(10):878-83. doi: 10.1016/j.cub.2013.04.001. Epub 2013 May 2. PMID 23643837
- [Background] Carpenter MJ, Saladin ME, Larowe SD, McClure EA, Simonian S, Upadhyaya HP, Gray KM. Craving, cue reactivity, and stimulus control among early-stage young smokers: effects of smoking intensity and gender. Nicotine Tob Res. 2014 Feb;16(2):208-15. doi: 10.1093/ntr/ntt147. Epub 2013 Sep 16. PMID 24042699